CLINICAL TRIAL: NCT07104708
Title: Effects of Systematic Exercise Training on Core Symptoms, Executive Function and Brain Function in Children With ASD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chen Li (Other)
Collaborators: Gansu Provincial Maternal and Child Health Care Hospital (Other)
Responsible Party: Sponsor-Investigator, Chen Li, Professor, Director, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SETA
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder
Keywords: executive function; brain function; exercise training; Autism spectrum disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The children are randomly divided into a intervention group and a control group. On the basis of the basic ASD rehabilitation training, the children will be trained for 12 weeks (5 days/week, 60 minutes/day). The intervention group received systematic exercise training (the Child-Parent- Trainer exercise program), while the control group received regular physical training courses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group received systematic exercise training (the Child-Parent- Trainer exercise program) for 12 weeks (5 days/week, 60 minutes/day).
  Interventions: Procedure: The Child-Parent- Trainer exercise program
- Control group (Active Comparator): The control group received regular physical training courses for 12 weeks (5 days/week, 60 minutes/day).
  Interventions: Procedure: The regular physical training

INTERVENTIONS:
Procedure: The Child-Parent- Trainer exercise program — The Child-Parent-Trainer exercise program is a 12-week exercise training program, which is based on the sensory and cognitive needs of children with ASD, multiple game forms are integrated to form a multi-sensory intervention model. The exercise program is developed according to the types of exercise recommended in the Exercise Guidelines for Preschool Children of China, including the development of basic motor skills, such as physical movement, posture control, object control; development of important physical qualities, such as agility, balance, coordination. The training program for different age group consists of physical movement items, object control items and limb coordination items. The exercise intensity is moderate.
  Arms: Intervention group
Procedure: The regular physical training — The regular physical training courses will last for 12 weeks. It is training in motor skills and fine motor skills. The items include passing the ball, lifting small dumbbells, running, handicrafts, etc. There is no requirement for the intensity of the exercise.
  Arms: Control group

SUMMARY:
Studies have shown that children with ASD simultaneously have deficits in overall executive function and impairments in basic motor skills, which have a negative impact on cognitive and social all-round development. In recent years, intervention measures for the motor skills of children with ASD have gradually developed. However, based on the existing literature, there is still a lack of recommendations for sports training at present. The sustained effect of exercise intervention training on the core symptoms of ASD remains unclear. In terms of executive function, there are relatively few studies on the executive function of preschool children. The impact of motor training on working memory in school-aged children is still inconsistent. Furthermore, the connection characteristics of different brain regions in children with ASD after physical training remain unclear. This study will include 70 children with ASD aged 3 to 9 years for a multicenter randomized controlled trial (RCT). These children will be randomly assigned to the intervention group (Child-Parent-Trainer program) and the control group (regular physical education program) for 12 weeks, 5 days/week, 60 minutes/day training. Children's core symptoms, executive function, child/family quality of life, and functional near-infrared spectroscopy (fNIRS) were assessed at baseline (training weeks 0) and endpoints (training weeks 13 and 17), respectively. To verify the improvement effect of this exercise program on the autism severity, core symptoms and executive functions of children with ASD, as well as its impact on family quality of life. Furthermore, through fNIRS for monitoring changes in brain function, the potential neural physiological mechanisms will be explored.

DETAILED DESCRIPTION:
1. Procedures. The children in the group are randomly divided into a intervention group and a control group. The children will be trained for 12 weeks (5 days/week, 60 minutes/day) and the children will be evaluated for the severity of autism, core symptoms, executive function, child/family quality of life, and fNIRS at training weeks 0, 13, and 17, respectively.
2. Demographic questionnaire and clinical data. The demographic questionnaire is completed by the child's primary caregiver, detailing child's name, gender, date of birth, height, weight, heart rate. Clinical data will be ascertained from the medical records, including information about DSM-5 diagnosis and comorbid conditions.
3. Sample size. This study is a randomized controlled trial. The proposed sample size is based on using the sample size formula, which compares the two sample means, . Where, tα is the standard normal difference corresponding to the level, taking α=0.05 and tα=1.96; tβ is the u value corresponding to the probability β of type II error, taking β=0.10 and tβ=1.28; σ is the estimate of the population standard deviation; δ is the allowable error, the difference between two population means. According to literature review, taking the adjustment ability in executive function as the main observation index, it is calculated that δ/σ =0.84. The sample size of intervention group and control group was 30 children, respectively. Considering the sample loss rate of 15%, the two groups are finally determined to be 35 children respectively.
4. Statistical analysis. SPSS 25.0 software (SPSS Inc) was used for statistical analysis for the scale data, including core symptoms and executive function, and the data were expressed as (M±SD). The scales scores and demographic variables of both groups of children will be compared using independent samples t-tests. Differences between baseline and 1 week and 1 month after exercise will be analysed using a repeated measures F-test. All statistical analyses were conducted with a statistical threshold P-value of <0.05. The data collected through fNIRS will be performed via NirSpark analysis software. The general linear model (GLM) will be applied to integrate task effects and assess activation in relevant brain regions. To analyze the rsFC of brain in children with ASD before and after the exercise intervention, the FC_NIRS toolbox is used.
5. Ethical matters and data protection. The patients participated in the study will sign the informed consent (obtained from the guardian). And this study was approved by the local ethics committee. Patient's name will be abbreviated and the research data will be assigned a code then to provide to the researcher. The authorization from parents on the patient's health information remains valid until the study is completed. After that, researchers will delete private information from the study record.

ELIGIBILITY:
Inclusion Criteria:

* Age: 3-9 years old.
* Meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnostic criteria for ASD, And hold a certificate of ASD diagnosis issued by a Tertiary A hospital.
* Borderline/normal intelligence or mild intellectual disability.
* No serious behavior or emotional problems.
* Able to simply ask and answer questions.
* Be able to proactively express the need to use the toilet.
* There are no physical impairments that affected participation in physical activities, and participants are able to cooperate to complete the intervention.
* Informed parental consent.

Exclusion Criteria:

* Vision/ hearing disorders, schizophrenia, emotional disorders, mental retardation, Rett syndrome and other developmental disorders.
* Medical conditions that limit the ability to be physically active, such as asthma, epilepsy, heart disease, and the acute phase after a fracture.
* History of head trauma, physical disability, major organ disease, or severe musculoskeletal injury in the past two years.
* Those who have participated in physical exercise regularly within the last 6 months.
* Participants who changed treatment intervention midway after inclusion.
* Unable to cooperate with persistent completion of intervention.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
The changes in degree of ASD disorder by Autism Diagnostic Observation Schedule-2 | Training weeks 0, 13, and 17.
  The changes in degree of ASD disorder by Autism Diagnostic Observation Schedule-2 Description: The Autism Diagnostic Observation Schedule-2 (ADOS-2) is adopted to assess the changes in the degree of ASD disorder. The Autism Diagnostic Observation Schedule-2 (ADOS-2) is a standardized observational assessment. The assessment includes abilities in four areas: social interaction, stereotypical behavior, verbal communication, emotion, and abnormal behavior. Children in the our study were administered a module 1 for children with little or no phrase speech or Module 2, for children who use phrase speech but are not yet fluent. Standardized ADOS scores in the domains of social affect (SA) and restricted repetitive behaviors (RRB) were calculated as indicators of ASD severity.
The changes in degree of ASD disorder by Childhood Autism Rating Scale (CARS) | Training weeks 0, 13, and 17.
  The Childhood Autism Rating Scale (CARS) are adopted to assess the changes in the degree of ASD disorder. The Childhood Autism Rating Scale (CARS) serves as an assessment indicator for the improvement of ASD symptoms. The scale consists of 15 items including relationship with people, imitation, emotional response, etc. The evaluation criteria for therapeutic effect are as follows: a CARS score reduction of less than or equal to 10 is considered effective, a CARS score reduction of 5 to 9 is considered effective, and a score reduction of less than 5 is considered ineffective.
The changes of executive functions | Training weeks 0, 13, and 17.
  The preschool BRIEF is consisted of 63 entries and divided into 5 factors and 3 dimensions. The 5 factors are inhibition, conversion, affective control, working memory, and organizational planning. The 3 dimensions are the inhibitory self-regulation index (including inhibition and affective control), cognitive flexibility index (including conversion and affective control) and metacognitive index (including working memory and organizational planning). School-age children BRIEF, consisting of 86 entries, is divided into 2 dimensions: behavior management index (including 3 factors of inhibition, conversion and emotional control) and metacognitive function index (including 5 factors of task initiation, working memory, planning, organization and monitoring). The higher the score, the more impaired the executive function. We examine the score of BRIEF to reflect changes in executive function before and after training.
The changes of brain function detection indicators | Training weeks 0, 13, and 17.
  We monitor cerebral hemodynamic changes through the fNIRS device. The Go/No-Go paradigm task was performed on children over 4 years old. This paradigm consists of two main parts, GO and GO /No-Go. During the GO task, participants are shown pictures of two animals (a giraffe and a lion) and instructed to quickly press the space bar when they see an animal picture. During the GO /No-Go task, pictures of two animals (a tiger and an elephant) are shown at random, and children are asked to quickly press the space bar when they see an elephant. To record correct rate and response time for analysis. All the subjects will undergo resting-state functional connectivity tests. We will compare the differences in fNIRS features before and after training.

SECONDARY OUTCOMES:
The changes of children's life quality by Child Eating Behavior Questionnaire (CEBQ) | Training weeks 0, 13, and 17.
  The dietary Behavior status of children was evaluated through the Child Eating Behavior Questionnaire (CEBQ). It includes 8 subscales such as food response, emotional overeating, and food preferences, covering 35 items. The answer score ranges from 1 to 5. If at least 80% of the items have been completed, the average value of each sub-scale will be calculated.
The changes of children's life quality by Children's Sleep Habits Questionnaire (CSHQ) | Training weeks 0, 13, and 17.
  The children's sleep habits questionnaire includes eight behaviors such as pre-sleep resistance, delayed sleep initiation, and sleep duration. A total score greater than 41 points indicates the presence of sleep disorders.
The changes of parents' life quality by Parenting Stress Index (PSI) | Training weeks 0, 13, and 17.
  The Parenting Stress Index was used to assess the mental stress that parents experience during the process of raising children. This scale consists of 36 items and covers 3 dimensions, including parenting distress, dysfunctional parent-child interaction, and children in difficulty. It is scored on a 5-point scale, with a higher score indicating greater parenting pressure. People with a total score of ≥P90 are considered to be under high pressure.
The changes in heart rate | At exercise training.
  Heart rate (or pulse rate) is the frequency of the heartbeat measured by the number of contractions (beats) of the heart per minute (bpm). When the children are doing aerobic exercise, we monitor the changes of heart rate and analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Li Chen, doctor, Study Director — Children's Hospital of Chongqing Medical University; yu T Li, Doctor, Study Chair — Children's Hospital of Chongqing Medical University
Locations (1):
- Growth, Development and Mental health of Children and Adolescence Center, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data is confidential during the study.

REFERENCES:
- [Result] Lord C, Elsabbagh M, Baird G, Veenstra-Vanderweele J. Autism spectrum disorder. Lancet. 2018 Aug 11;392(10146):508-520. doi: 10.1016/S0140-6736(18)31129-2. Epub 2018 Aug 2. PMID 30078460
- [Result] Xu G, Strathearn L, Liu B, O'Brien M, Kopelman TG, Zhu J, Snetselaar LG, Bao W. Prevalence and Treatment Patterns of Autism Spectrum Disorder in the United States, 2016. JAMA Pediatr. 2019 Feb 1;173(2):153-159. doi: 10.1001/jamapediatrics.2018.4208. PMID 30508021
- [Result] Demetriou EA, Lampit A, Quintana DS, Naismith SL, Song YJC, Pye JE, Hickie I, Guastella AJ. Autism spectrum disorders: a meta-analysis of executive function. Mol Psychiatry. 2018 May;23(5):1198-1204. doi: 10.1038/mp.2017.75. Epub 2017 Apr 25. PMID 28439105
- [Result] Lippi G, Mattiuzzi C, Sanchis-Gomar F. Updated overview on interplay between physical exercise, neurotrophins, and cognitive function in humans. J Sport Health Sci. 2020 Jan;9(1):74-81. doi: 10.1016/j.jshs.2019.07.012. Epub 2019 Sep 6. PMID 31921482
- [Result] Zampella CJ, Wang LAL, Haley M, Hutchinson AG, de Marchena A. Motor Skill Differences in Autism Spectrum Disorder: a Clinically Focused Review. Curr Psychiatry Rep. 2021 Aug 13;23(10):64. doi: 10.1007/s11920-021-01280-6. PMID 34387753
- [Result] Chan JS, Deng K, Yan JH. The effectiveness of physical activity interventions on communication and social functioning in autistic children and adolescents: A meta-analysis of controlled trials. Autism. 2021 May;25(4):874-886. doi: 10.1177/1362361320977645. Epub 2020 Dec 11. PMID 33307759
- [Result] Sandbank M, Bottema-Beutel K, Woynaroski T. Intervention Recommendations for Children With Autism in Light of a Changing Evidence Base. JAMA Pediatr. 2021 Apr 1;175(4):341-342. doi: 10.1001/jamapediatrics.2020.4730. No abstract available. PMID 33165523
- [Result] Jia M, Zhang J, Pan J, Hu F, Zhu Z. Benefits of exercise for children and adolescents with autism spectrum disorder: a systematic review and meta-analysis. Front Psychiatry. 2024 Oct 7;15:1462601. doi: 10.3389/fpsyt.2024.1462601. eCollection 2024. PMID 39435130
- [Result] Tao R, Yang Y, Wilson M, Chang JR, Liu C, Sit CHP. Comparative effectiveness of physical activity interventions on cognitive functions in children and adolescents with Neurodevelopmental Disorders: a systematic review and network meta-analysis of randomized controlled trials. Int J Behav Nutr Phys Act. 2025 Jan 13;22(1):6. doi: 10.1186/s12966-024-01702-7. PMID 39806448
- [Result] Chan AS, Sze SL, Siu NY, Lau EM, Cheung MC. A chinese mind-body exercise improves self-control of children with autism: a randomized controlled trial. PLoS One. 2013 Jul 10;8(7):e68184. doi: 10.1371/journal.pone.0068184. Print 2013. PMID 23874533
- [Result] Toscano CVA, Ferreira JP, Quinaud RT, Silva KMN, Carvalho HM, Gaspar JM. Exercise improves the social and behavioral skills of children and adolescent with autism spectrum disorders. Front Psychiatry. 2022 Dec 22;13:1027799. doi: 10.3389/fpsyt.2022.1027799. eCollection 2022. PMID 36620673
- [Result] Grospretre S, Ruffino C, Derguy C, Gueugneau N. Sport and Autism: What Do We Know so Far? A Review. Sports Med Open. 2024 Oct 3;10(1):107. doi: 10.1186/s40798-024-00765-x. PMID 39361117
- [Result] Zhang F, Roeyers H. Exploring brain functions in autism spectrum disorder: A systematic review on functional near-infrared spectroscopy (fNIRS) studies. Int J Psychophysiol. 2019 Mar;137:41-53. doi: 10.1016/j.ijpsycho.2019.01.003. Epub 2019 Jan 19. PMID 30664885
- [Result] Mazzoni A, Grove R, Eapen V, Lenroot RK, Bruggemann J. The promise of functional near-infrared spectroscopy in autism research: What do we know and where do we go? Soc Neurosci. 2019 Oct;14(5):505-518. doi: 10.1080/17470919.2018.1497701. Epub 2018 Jul 21. PMID 29985114
- [Result] Deng J, Lei T, Du X. Effects of sensory integration training on balance function and executive function in children with autism spectrum disorder: evidence from Footscan and fNIRS. Front Psychol. 2023 Oct 25;14:1269462. doi: 10.3389/fpsyg.2023.1269462. eCollection 2023. PMID 37946875
- [Result] Chen H, Liang Q, Wang B, Liu H, Dong G, Li K. Sports game intervention aids executive function enhancement in children with autism - An fNIRS study. Neurosci Lett. 2024 Feb 6;822:137647. doi: 10.1016/j.neulet.2024.137647. Epub 2024 Jan 17. PMID 38242348
- [Result] Yeung MK. An optical window into brain function in children and adolescents: A systematic review of functional near-infrared spectroscopy studies. Neuroimage. 2021 Feb 15;227:117672. doi: 10.1016/j.neuroimage.2020.117672. Epub 2020 Dec 24. PMID 33359349
- [Result] Xu L, Hua Q, Yu J, Li J. Classification of autism spectrum disorder based on sample entropy of spontaneous functional near infra-red spectroscopy signal. Clin Neurophysiol. 2020 Jun;131(6):1365-1374. doi: 10.1016/j.clinph.2019.12.400. Epub 2020 Jan 13. PMID 32311592
- [Result] Eng CM, Pocsai M, Fulton VE, Moron SP, Thiessen ED, Fisher AV. Longitudinal investigation of executive function development employing task-based, teacher reports, and fNIRS multimethodology in 4- to 5-year-old children. Dev Sci. 2022 Nov;25(6):e13328. doi: 10.1111/desc.13328. Epub 2022 Oct 21. PMID 36221252